CLINICAL TRIAL: NCT06561685
Title: An Open-label, Multicenter Study of LY4050784, a Selective SMARCA2/BRM Inhibitor, in Advanced Solid Tumor Malignancies With SMARCA4/BRG1 Alterations
Brief Title: A Study of LY4050784 in Participants With Advanced or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 27191; J5M-OX-JOXA (Other: Eli Lilly and Company)
Record Dates: First submitted 2024-08-16; First posted 2024-08-20 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Metastatic Solid Tumor; Advanced Solid Tumor; Non-small Cell Lung Cancer; SMARCA4-Deficient Tumor
Keywords: SMARCA2; SMARCA4; Lung cancer; BRM; BRG1; Adenocarcinoma; Squamous cell carcinoma; Targeted therapy
MeSH Terms: conditions — Neoplasm Metastasis; Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Adenocarcinoma; Carcinoma, Squamous Cell | interventions — pembrolizumab; Cisplatin; Carboplatin; Pemetrexed; Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- LY4050784 (Phase 1a - Dose Escalation) (Experimental): Escalating doses of LY4050784 administered orally.
  Interventions: Drug: LY4050784
- LY4050784 (Phase 1b - Dose Optimization/Part A) (Experimental): Comparing 2 or more doses (evaluated during dose escalation) of LY4050784 administered orally.
  Interventions: Drug: LY4050784
- LY4050784 (Phase 1b - Dose Expansion/Part B) (Experimental): LY4050784 administered orally.
  Interventions: Drug: LY4050784
- LY4050784 (Phase 1b - Dose Expansion/Part C) Cohort C1 (Experimental): LY4050784 administered orally in combination in combination with pembrolizumab administered IV in 21-day cycles. Participants may continue to receive treatment until discontinuation criteria are met.
  Interventions: Drug: LY4050784; Drug: Pembrolizumab
- LY4050784 (Phase 1b - Dose Expansion/Part C) Cohort C2a (Experimental): LY4050784 administered orally in combination in combination with pembrolizumab, pemetrexed, and platinum (cisplatin or carboplatin) administered IV in 21-day cycles. Participants may continue to receive treatment until discontinuation criteria are met.
  Interventions: Drug: LY4050784; Drug: Pembrolizumab; Drug: Cisplatin; Drug: Carboplatin; Drug: Pemetrexed
- LY4050784 (Phase 1b - Dose Expansion/Part C) Cohort C2b (Experimental): LY4050784 administered orally in combination in combination with pembrolizumab, paclitaxel/nab-paclitaxel and carboplatin administered IV in 21-day cycles. Participants may continue to receive treatment until discontinuation criteria are met.
  Interventions: Drug: LY4050784; Drug: Pembrolizumab; Drug: Carboplatin; Drug: Paclitaxel; Drug: Nab paclitaxel

INTERVENTIONS:
Drug: LY4050784 — Oral
Drug: Pembrolizumab — Administered IV.
  Arms: LY4050784 (Phase 1b - Dose Expansion/Part C) Cohort C1; LY4050784 (Phase 1b - Dose Expansion/Part C) Cohort C2a; LY4050784 (Phase 1b - Dose Expansion/Part C) Cohort C2b
Drug: Cisplatin — Administered IV.
  Arms: LY4050784 (Phase 1b - Dose Expansion/Part C) Cohort C2a
Drug: Carboplatin — Administered IV.
  Arms: LY4050784 (Phase 1b - Dose Expansion/Part C) Cohort C2a; LY4050784 (Phase 1b - Dose Expansion/Part C) Cohort C2b
Drug: Pemetrexed — Administered IV.
  Arms: LY4050784 (Phase 1b - Dose Expansion/Part C) Cohort C2a
Drug: Paclitaxel — Administered IV.
  Arms: LY4050784 (Phase 1b - Dose Expansion/Part C) Cohort C2b
Drug: Nab paclitaxel — Administered IV.
  Arms: LY4050784 (Phase 1b - Dose Expansion/Part C) Cohort C2b

SUMMARY:
The main purpose of this study is to find out whether the study drug, LY4050784, is safe, tolerable and effective in participants alone or in combination with other anticancer agents. In addition, with locally advanced or metastatic solid tumors with a BRG1 (Brahma-related gene 1, also known as SMARCA4) alteration who have previously received, do not qualify for, or are refusing standard of care treatments, or there is no standard therapy available for the disease. The study is conducted in two parts - phase Ia (dose-escalation) and phase Ib (dose-optimization, dose-expansion). The study will last up to approximately 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Have one of the following locally advanced or metastatic solid tumor malignancy with SMARCA4 (BRG1) alteration:

  * Phase 1a dose escalation: Presence of any alteration in SMARCA4 (BRG1)
  * Phase 1b expansion: Part A: Non-small Cell Lung Cancer (NSCLC) that is locally advanced and not suitable for definitive locoregional therapy, or metastatic with presence of a known or likely loss of function alteration in SMARCA4 (BRG1) or loss of protein expression.
  * Phase 1b expansion: Part B: Any tumor type (other than NSCLC) that has the presence of a known or likely loss of function alteration in SMARCA4 (BRG1) or loss of protein expression.
  * Phase 1b expansion: Part C: Non-small Cell Lung Cancer (NSCLC) that is locally advanced and not suitable for definitive locoregional therapy, or metastatic with presence of a known or likely loss of function alteration in SMARCA4 (BRG1) or loss of protein expression.
* Prior Systemic Therapy Criteria:

  * Phase 1a dose escalation and Phase 1b (Part B): Participants who received all standard therapies for which the individual was deemed to be an appropriate candidate by the treating Investigator; or the individual is refusing the remaining most appropriate standard of care treatment; or there is no standard therapy available for the disease.
  * Phase 1b expansion (Part A): Participants must have received at least one line of therapy for advanced or metastatic disease.
  * Phase 1b expansion (Part C): Participants may be treatment naïve or have received therapy for advanced or metastatic disease
* Measurability of disease

  * Phase 1a dose escalation (excluding backfill): measurable or non-measurable disease as defined by Response Evaluation Criteria in Solid Tumors v1.1 (RECIST v1.1)
  * Phase 1a backfill and Phase 1b expansion: Measurable disease required as defined by RECIST v1.1
* Have an Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1

Exclusion Criteria:

* Participants with known or likely loss of function alteration of SMARCA2 (BRM) or malignancy with known association with SMARCA2 (BRM) alterations
* Prior exposure to SMARCA2 (BRM) inhibitor(s) and/or degrader(s) (prior exposure may be permitted for dose escalation)
* Participants with known or suspected history of untreated or uncontrolled central nervous system (CNS) involvement
* Participants with history of increased risk of prolonged QT or significant arrythmia
* Significant cardiovascular disease
* Participants with active and/or treated for an additional primary malignancy within 2 years prior to enrolment
* Participants who are pregnant, breastfeeding or plan to breastfeed or expecting to conceive or father children during study or within 6 months after the last dose of study intervention
* Participants with history of active autoimmune diseases, history of allogenic stem cell/organ transplant or compromised immune system within past 2 years (Part C only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2024-09-19 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Phase Ia: Number of Participants with One or More Treatment Emergent Adverse Events (TEAEs), Serious Adverse Event(s) (SAEs), and Adverse Event(s) (AEs) | Up to Approximately 48 Months or 4 Years
  A summary of TEAEs, SAEs, and AEs regardless of causality, will be reported in the Reported Adverse Events module
Phase 1a: To determine the maximum tolerated dose (MTD)/recommended phase 2 dose (RP2D) of LY4050784 | Up to Approximately 48 Months or 4 Years
  Number of participants with dose-limiting toxicities (DLTs)
Phase 1b: To assess the antitumor activity of LY4050784 Monotherapy: Overall response rate (ORR) | Up to Approximately 48 Months or 4 Years
  ORR per investigator assessed Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST 1.1)
Phase 1b (Dose optimization only): To confirm the RP2D/optimal dose based on safety and efficacy of LY4050784 | Up to Approximately 48 Months or 4 Years
  A summary of TEAEs, SAEs, and AEs regardless of causality, will be reported in the Reported Adverse Events module, ORR and Duration of Response (DOR) per Investigator
Phase 1b (Combination cohorts/Part C): To assess the safety and tolerability of LY4050784 when administered in combination with other anticancer agents | Up to Approximately 48 Months or 4 Years
  A summary of TEAEs, SAEs, and AEs regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
To characterize the pharmacokinetics (PK) properties of LY4050784: Maximum Concentration (Cmax) | Cycle 1 (Day 8)
  PK: Cmax of LY4050784
To characterize the PK properties of LY4050784: Time to Maximum Concentration (Tmax) | Cycle 1 (Day 8)
  PK: Tmax of LY4050784
To characterize the PK properties of LY4050784: Area under the concentration versus time curve (AUC) | Cycle 1 (Day 8)
  PK: AUC of LY4050784
Phase Ia: To evaluate the preliminary antitumor activity of LY4050784: Overall response rate (ORR) | Up to Approximately 48 Months or 4 Years
  ORR per investigator assessed Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST 1.1)
To evaluate the preliminary antitumor activity of LY4050784: Duration of response (DOR) | Up to Approximately 48 Months or 4 Years
  DOR per investigator assessed RECIST 1.1
To evaluate the preliminary antitumor activity of LY4050784: Time to response (TTR) | Up to Approximately 48 Months or 4 Years
  TTR per investigator assessed RECIST 1.1
To evaluate the preliminary antitumor activity of LY4050784: Disease control rate (DCR) | Up to Approximately 48 Months or 4 Years
  DCR per investigator assessed RECIST 1.1
To evaluate the preliminary antitumor activity of LY4050784: Progression free survival (PFS) | Up to Approximately 48 Months or 4 Years
  PFS per investigator assessed RECIST 1.1
To evaluate the PK properties of LY4050784 in combination cohorts: Maximum Concentration (Cmax) PK: Cmax of LY4050784 | Cycle 1 (Day 8)
To evaluate the PK properties of LY4050784 in combination cohorts: Time to Maximum Concentration (Tmax) PK: Tmax of LY4050784 | Cycle 1 (Day 8)
To evaluate the PK properties of LY4050784 in combination cohorts: Area under the concentration versus time curve (AUC) | Cycle 1 (Day 8)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (33):
- United States (17):
  - UCLA, Santa Monica, California
  - University of Colorado Health Hospital, Aurora, Colorado
  - Sarah Cannon Research Institute at HealthOne, Denver, Colorado
  - Florida Cancer Specialists ORLANDO/DDU, Lake Mary, Florida
  - University of Miami, Miami, Florida
  - University of Chicago, New Lenox, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Ohio State University Hospital, Columbus, Ohio
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - SCRI Oncology Partners, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - USO-Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- France (3):
  - Institut Bergonie, Bordeaux
  - Institut Curie, Paris
  - Institut Gustave Roussy-Gustave Roussy Cancer Center -DITEP, Villejuif
- Germany (3):
  - Charite-Universitatsmedizin Berlin, Berlin
  - Universitaetsklinikum Essen, Essen
  - Krankenhaus Nordwest, Frankfurt am Main
- Japan (5):
  - National Cancer Center Hospital, Chūōku
  - National Cancer Center Hospital East, Kashiwa
  - The Cancer Institute Hospital of JFCR, Kōtō City
  - Shizuoka Cancer Center, Nagaizumi-cho,Sunto-gun
  - Aichi Cancer Center Hospital, Nagoya
- South Korea (3):
  - National Cancer Center, Ilsandong-gu
  - Severance Hospital, Yonsei University Health System, Seoul
  - The Catholic University of Korea, St. Vincent's Hospital, Suwon
- Spain (2):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - South Texas Accelerated Research Therapeutics (START) Madrid - Hospital Fundacion Jimenez Diaz, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Study of LY4050784 in Participants With Advanced or Metastatic Solid Tumors — https://trials.lilly.com/en-US/trial/528616